CLINICAL TRIAL: NCT03014791
Title: Influence of Age, Weight and Ethnic Background on Blood Pressure: AWE Study
Brief Title: Influence of Age, Weight and Ethnic Background on Blood Pressure
Acronym: AWE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Collaborators: University of Cambridge (Other)
Responsible Party: Principal Investigator, Carmel McEniery, Senior Research Associate, Cambridge University Hospitals NHS Foundation Trust
Other Study IDs: AWE
Record Dates: First submitted 2017-01-06; First posted 2017-01-09 (Estimated); Last update posted 2022-08-23 (Actual); Status verified 2022-08

CONDITIONS: Cardiovascular Diseases; Vascular Diseases; Hypertension
Keywords: Epidemiology; Ethnicity; Age; Weight; Hypertensive; Cardiac Output; Peripheral Vascular Resistance; Arterial Stiffness; Healthy Volunteers; Endothelial function; Arterial Structure; Left ventricular mass/function
MeSH Terms: conditions — Cardiovascular Diseases; Vascular Diseases; Hypertension; Body Weight | interventions — Blood Pressure; Vascular Stiffness; Cardiac Output; Ventilation; Blood Specimen Collection; Urine Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — During the study, the blood and urine samples will be stored by the research team at the department of Experimental Medicine and Immunotherapeutics, Division of Cardiovascular Medicine under the responsibility of the CI who will ensure the security and confidentiality of the stored material. These samples will not be accessible to any investigator outside the research team. A small aliquot of the participant's blood and urine sample will be stored at approximately -80 degrees Celsius for future analyses. All samples taken during this study will be made anonymous. Samples obtained during this study will be used for future ethically approved studies. Participants will be made aware of this in the participant information sheet prior to the process of written informed consent.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Healthy Volunteers: No IMP to be administered, only challenge agents as part of the physiological assessments.
  Large artery endothelial function:
  * Glyceryl trinitrate 500 μg (Sublingual administration to stimulate endothelium-independent vasodilatation)
  * Salbutamol 2 x 200 μg (Administered by spacer device to stimulate endothelium-dependent vasodilatation)
  Forearm blood flow
  * Acetylcholine: 7.5μg/min, 15μg/min and 30μg/min (Intra-arterial administration via brachial artery to stimulate endothelium-dependent vasodilatation)
  * Sodium nitroprusside: 3μg/min, 10μg/min (Intra-arterial administration via brachial artery to stimulate endothelium-independent vasodilatation)
  * LNMMA: 2μmol/min, 4μmol/min (Intra-arterial administration via brachial artery to block basal nitric oxide production)
  Interventions: Other: Brief lifestyle/medical history questionnaire; Other: Anthropometric measures; Other: Blood pressure and arterial stiffness; Other: Cardiac output and lung function; Other: Heart rate variability; Other: Blood sample & spot urine sample; Other: 24 hour ambulatory blood pressure monitor; Other: 24 hour urine collection; Other: Echocardiograph: Left ventricular mass; Other: Large artery structure: Carotid intima-media thickness; Other: Small artery structure: Minimum forearm vascular resistance; Other: Large artery endothelial function; Other: Small artery endothelial function: Forearm blood flow; Other: Dundee step test; Other: Detailed haemodynamic response to submaximal exercise; Other: Cardiopulmonary fitness: Maximum oxygen consumption; Other: Haemodynamic response to mental stress; Other: Small artery dilatory function: Forearm blood flow
- Hypertensive Patients (Case-control): No IMP to be administered, only challenge agents as part of the physiological assessments.
  Large artery endothelial function:
  * Glyceryl trinitrate 500 μg (Sublingual administration to stimulate endothelium-independent vasodilatation)
  * Salbutamol 2 x 200 μg (Administered by spacer device to stimulate endothelium-dependent vasodilatation)
  Forearm blood flow
  * Acetylcholine: 7.5μg/min, 15μg/min (Intra-arterial administration via brachial artery to stimulate endothelium-dependent vasodilatation)
  * Sodium nitroprusside: 3μg/min, 10μg/min (Intra-arterial administration via brachial artery to stimulate endothelium-independent vasodilatation)
  * LNMMA: 2μmol/min, 4μmol/min (Intra-arterial administration via brachial artery to block basal nitric oxide production)
  Interventions: Other: Brief lifestyle/medical history questionnaire; Other: Anthropometric measures; Other: Blood pressure and arterial stiffness; Other: Cardiac output and lung function; Other: Heart rate variability; Other: Blood sample & spot urine sample; Other: 24 hour ambulatory blood pressure monitor; Other: 24 hour urine collection; Other: Echocardiograph: Left ventricular mass; Other: Large artery structure: Carotid intima-media thickness; Other: Small artery structure: Minimum forearm vascular resistance; Other: Large artery endothelial function; Other: Small artery endothelial function: Forearm blood flow; Other: Dundee step test; Other: Detailed haemodynamic response to submaximal exercise; Other: Cardiopulmonary fitness: Maximum oxygen consumption; Other: Haemodynamic response to mental stress; Other: Small artery dilatory function: Forearm blood flow
- Hypertensive Patients (Cross-sectional): No IMP to be administered, only challenge agents as part of the physiological assessments.
  Large artery endothelial function:
  Same challenge agents as healthy volunteer and hypertensive patient (Case-control) arms
  Forearm blood flow Same challenge agents as healthy volunteer and hypertensive patient (Case-control) arms
  Recruited from community-based cohort studies - CLEAREST and ACCT
  Equal recruitment across the following parameters:
  * Age: 3 groups <30, 30-60, >60 years
  * Gender
  * BMI: 3 groups <25, 25-30, >30 Kg/m2
  Interventions: Other: Brief lifestyle/medical history questionnaire; Other: Anthropometric measures; Other: Blood pressure and arterial stiffness; Other: Cardiac output and lung function; Other: Heart rate variability; Other: Blood sample & spot urine sample; Other: 24 hour ambulatory blood pressure monitor; Other: 24 hour urine collection; Other: Echocardiograph: Left ventricular mass; Other: Large artery structure: Carotid intima-media thickness; Other: Small artery structure: Minimum forearm vascular resistance; Other: Large artery endothelial function; Other: Small artery endothelial function: Forearm blood flow; Other: Dundee step test; Other: Detailed haemodynamic response to submaximal exercise; Other: Cardiopulmonary fitness: Maximum oxygen consumption; Other: Haemodynamic response to mental stress; Other: Small artery dilatory function: Forearm blood flow

INTERVENTIONS:
Other: Brief lifestyle/medical history questionnaire — Core Measurement
Other: Anthropometric measures — Core Measurement
Other: Blood pressure and arterial stiffness — Core Measurement
Other: Cardiac output and lung function — Core Measurement
Other: Heart rate variability — Core Measurement
Other: Blood sample & spot urine sample — Core Measurement
Other: 24 hour ambulatory blood pressure monitor — Detailed Measurement (Optional for participants).
Other: 24 hour urine collection — Detailed Measurement (Optional for participants).
Other: Echocardiograph: Left ventricular mass — Detailed Measurement (Optional for participants).
Other: Large artery structure: Carotid intima-media thickness — Detailed Measurement (Optional for participants).
Other: Small artery structure: Minimum forearm vascular resistance — Detailed Measurement (Optional for participants).
Other: Large artery endothelial function — Flow- and salbutamol-mediated vasodilatation Detailed Measurement (Optional for participants).
Other: Small artery endothelial function: Forearm blood flow — Detailed Measurement (Optional for participants).
Other: Dundee step test — Systolic blood pressure response to submaximal exercise Detailed Measurement (Optional for participants).
Other: Detailed haemodynamic response to submaximal exercise — Detailed Measurement (Optional for participants).
Other: Cardiopulmonary fitness: Maximum oxygen consumption — Detailed Measurement (Optional for participants).
Other: Haemodynamic response to mental stress — Detailed Measurement (Optional for participants).
Other: Small artery dilatory function: Forearm blood flow — Detailed Measurement (Optional for participants).

SUMMARY:
Hypertension, also known as high blood pressure, is a chronic medical condition, in which the blood pressure is elevated. This is a common condition, which can lead to severe complications such as cardiovascular disease, heart attack, stroke and kidney disease, if not detected and treated early.

Accumulating evidence suggests that the incidence of hypertension varies according to age, ethnicity and obesity. In order to obtain an in-depth knowledge of the pathophysiological mechanisms of hypertension, we aim to investigate the haemodynamic and biochemical correlates of elevated blood pressure across the adult age-span, and determine the extent to which body size and ethnicity impact on these associations. We also wish to investigate the impact of hypertension on key target organs (end-organ damage). The primary objective of this study is to compare the mechanisms regulating blood pressure in hypertensive and non-hypertensive participants across the adult age span, and to assess the influence of body mass index and ethnic background on these mechanisms. Secondary objectives are to investigate the association between blood pressure and cardiovascular physiology across the adult age span at rest and during sub-maximal exercise and to investigate the impact of blood pressure haemodynamics on key organs including the arteries and heart by assessing end-organ damage such as endothelial function, arterial structure and left ventricular mass/function.

This study will be a combined case-control and cross-sectional study describing the procedures and time commitment required to investigate our scientific aims. This is a single centre study that will be conducted in a secondary care environment. Both male and females aged 18 and over and that are able provide informed consent will be considered for this study. People who are pregnant, currently receiving dialysis, illness with a life expectancy <1 year, current active malignancy and cannot provide informed consent are ineligible for this study. The study will be open for five years and each patient will complete a maximum of four visits in a 12 month period. Participants will complete a variety of non-invasive physiological assessments of their cardiovascular system and lung function. There will be some minimally invasive procedures completed, including a blood test and assessment of small artery endothelial function which involves insertion of a small needle under local anesthetic.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female, aged 18 or above
* Able to give informed consent and willing to participate

Exclusion Criteria:

* Pregnancy
* Current active malignancy
* Currently receiving dialysis
* Any illness with a life expectancy < 1 year
* Lack of written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Hypertensive patients for this study will be identified in a secondary care setting from hypertension clinics at Cambridge University Hospitals, from two on-going observational community-based cohort studies - CLEAREST and ACCT, in addition to potential participants (healthy volunteers) who respond to recruitment posters displayed around Cambridge University Hospitals and the University of Cambridge.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2017-02-21 (Actual); Primary Completion 2024-02 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Cardiac Output (Measured by the inert gas re-breathing technique L/Min) | 5 years
Peripheral vascular resistance (Calculated using Cardiac Output and Blood pressure data dynes/sec/cm^5 ) | 5 years
Pulse wave velocity (Measured by ECG-gated applanation tonometry meters/sec) | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Carmel McEniery, PhD, Principal Investigator — University of Cambridge
Locations (1):
- Vascular Research Clinic, Addenbrooke's Hospital, Cambridge, Cambridgeshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No